CLINICAL TRIAL: NCT01657825
Title: A Phase 1, Open-Label, Sequential Study of the Effect of Multiple Doses of Isavuconazole on the Pharmacokinetics of a Single Dose of Warfarin in Healthy Male Subjects
Brief Title: Drug Interaction Study of Isavuconazole and Warfarin in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Basilea Pharmaceutica International Ltd (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 9766-CL-0033
Record Dates: First submitted 2012-08-02; First posted 2012-08-06 (Estimated); Last update posted 2012-08-28 (Estimated); Status verified 2012-08

CONDITIONS: Pharmacokinetics of Isavuconazole; Pharmacokinetics of S- and R-warfarin; Pharmacodynamics of Warfarin; Healthy Volunteers
Keywords: isavuconazole; warfarin; Healthy Volunteers; BAL8557; Coumadin
MeSH Terms: interventions — isavuconazole; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Isavuconazole and warfarin (Experimental): Isavuconazole three times daily (TID) for 2 days followed by once daily (QD) dosing for 11 days and warfarin single doses on Days 1 and 20
  Interventions: Drug: Isavuconazole; Drug: Warfarin

INTERVENTIONS:
Drug: Isavuconazole — oral
  Other Names: BAL8557
Drug: Warfarin — oral
  Other Names: Coumadin

SUMMARY:
The purpose of this study is to assess the effect of multiple doses of isavuconazole on the pharmacokinetics (PK) of warfarin after single dose administration.

DETAILED DESCRIPTION:
Subjects will receive a single dose of warfarin on Day 1 followed by a 15 day wash-out period (time from warfarin dosing to isavuconazole dosing).

On Days 16 and 17, isavuconazole will be dosed three times daily (TID). TID doses will be administered 8 hours apart. On Days 18 through 28, isavuconazole will be administered once daily (QD). All subjects will be administered a single dose of warfarin on Day 20. A follow up visit will occur approximately 7 days after the last dose of isavuconazole. Blood samples for pharmacokinetics will be collected throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have BMI of 18 to 32 kg/m2 and a body weight of at least 45 kg
* Subjects must have normal laboratory values especially for ALT, AST, protein C and S, and prothrombin time

Exclusion Criteria:

* The subject has a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmia or torsade de pointes, structural heart disease, or family history of Long QT syndrome (suggested by sudden death of a close relative at a young age due to possible or probable cardiac causes)
* The subject has a positive result for hepatitis C antibodies or hepatitis B surface antigen at Screening or is known to be positive for human immunodeficiency virus (HIV)
* The subject has a known or suspected allergy to any of the components of the trial products or the azole class of compounds, or a history of multiple and/or severe allergies to drugs or foods (as judged by the investigator), or a history of severe anaphylactic reactions
* The subject is a smoker (any use of tobacco or nicotine containing products) within 6 months prior to Screening
* The subject has had treatment with prescription drugs or complementary and alternative medicines within 14 days prior to Day -1, or over-the-counter medications within 1 week prior to Day -1
* The subject has received an experimental agent within 30 days or 5 half-lives, whichever is longer prior to Day -1
* The subject has a recent history (within the last 2 years) of drug or alcohol abuse, as defined by the investigator, or a positive drug and/or alcohol screen

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Composite of Pharmacokinetic (PK) variables for S-warfarin (in plasma): AUCinf, AUClast, Cmax | Days 1 and 20, predose and at 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12,16, 24, 48, 72, 96, 120, 144, 168, and 216 hours postdose
  Area under the curve (AUC) from time 0 extrapolated to infinity (AUCinf), AUC from time of dosing to last quantifiable concentration (AUClast ), and maximum concentration (Cmax)

SECONDARY OUTCOMES:
Composite of PK variables for R-warfarin (in plasma): AUCinf, AUClast, Cmax | Days 1 and 20, predose and at 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12,16, 24, 48, 72, 96, 120, 144, 168, and 216 hours postdose
Composite of Pharmacokinetic (PK) variables for S-warfarin and R-warfarin (in plasma): tmax, Vz /F, CL/F, and t1/2 | Days 1 and 20, predose and at 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12,16, 24, 48, 72, 96, 120, 144, 168, and 216 hours postdose
  Time to attain Cmax (tmax) , apparent volume of distribution (Vz /F), apparent body clearance after oral dosing (CL/F), and apparent terminal elimination half-life (t1/2)
PK variable for isavuconazole (in plasma): trough concentration (Ctrough) | Days 18-20 and Days 22-27, predose and Day 28 predose and 24 hours post dose
Composite of PK variable for isavuconazole (in plasma): AUCtau , Cmax, and tmax | Day 19 predose and at 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 and 16 hours post dose; and Day 20, predose and at 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24, and 36 hours postdose
  AUC during the time interval between consecutive dosing (AUCtau)
Pharmacodynamic Variables: MAXINR, AUCINR, MAXPT, and AUCPT | Day 1 and Day 20 predose and at 6, 12, 24, 48, 72, 96, 168, and 216 hours post-warfarin-dose
  International Normalized Ratio (INR), Maximum observed change INR value (MAXINR), Area under the INR time curve from 0 to 216 hours (AUCINR), Maximum observed change in prothrombin time (PT)value (MAXPT), Area under the PT time curve from 0 to 216 hours (AUCPT)
Safety assessed by recording of adverse events, clinical laboratory evaluation, electrocardiograms (ECGs) physical examinations, and vital signs | Day 1 through Day 29, Day 35 ± 2

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (1):
- Spaulding Clinical, West Bend, Wisconsin, United States